CLINICAL TRIAL: NCT00832273
Title: Use of the Extracorporeal Liver Assist Device (ELAD®) In Patients With Liver Failure: Uncontrolled Treatment Protocol to Provide Expanded Access With Cost Recovery
Brief Title: Use of the ELAD® in Patients With Liver Failure to Provide Expanded Access With Cost Recovery
Status: No longer available | Type: Expanded Access
Sponsor: Vital Therapies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VTI-501
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Liver Failure
Keywords: Expanded access to ELAD® in patients with liver failure
MeSH Terms: conditions — Liver Failure

INTERVENTIONS:
Device: ELAD® — liver assist system

SUMMARY:
VTI had established other clinical protocols to study the effects of ELAD® plus standard therapy compared with standard therapy alone in patients with acute on chronic (AOCH) (VTI-201, VTI-206) and fulminant hepatic failure (FHF) (VTI-202) and acute alcoholic hepatitis (AAH). However, liver failure (LF) patients who do not qualify for other protocols may benefit from ELAD use. In order to accommodate physician requests for the use of ELAD in LF patients who do not qualify for open Protocols, without the need to resort to individual Emergency Use INDs for each case, VTI has developed a Treatment Protocol with Cost Recovery to provide for expanded access to ELAD for those with LF. This uncontrolled Treatment Protocol has been designed to provide expanded access to ELAD in subjects with LF while assuring that sufficient data are collected to adequately monitor ELAD safety when used in this setting at multiple centers in the United States.

DETAILED DESCRIPTION:
ELAD® therapy is designed to provide continuous liver support to a subject with compromised liver function, allowing time for the subject's native liver to regenerate to a healthy state, or to stabilize the subject until a suitable donor organ can be found for transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Weight ≥15 kg;
2. Age ≥10 and ≤70 years;
3. MELD score of ≥24;
4. Documented liver failure;
5. Subject or designated representative must be willing to sign an Informed Consent Form specific to this study and comply with study requirements.

Exclusion Criteria:

1. Cerebral Perfusion Pressure (CPP) as measured by an intracranial pressure (ICP) monitor.:

   1. Patients ≥ 18 yrs of age with Cerebral Perfusion Pressures ≤40 mm Hg for one hour or longer.
   2. Patients ≤18 yrs with CPP ≤35 mm Hg for one hour or longer.
2. Concomitant disease including chronic congestive heart failure, vascular disease, emphysema, AIDS, cancer, acute fatty-liver disease, hepatitis due to herpes virus, Wilson's disease, or Budd-Chiari syndrome;
3. Portal hypertension;
4. Liver dysfunction due to trauma;
5. Hemorrhage or irreversible brain death;
6. Platelet count <50,000/mm3 or reducing to <80,000/mm3 over a 72 hour period;
7. Mean Arterial Pressures (MAP) ≤50 mm Hg for one hour or longer as measured by an indwelling arterial line, OR; patients ≤18 years old and whose MAP is ≤40 mm Hg for one hour or longer;
8. Vasopressor support exceeding 1.0 µg/kg/min of an alpha-adrenergic agent for one hour or longer;
9. Clinical or radiographic evidence of stroke or intracerebral bleeding;
10. Seizures uncontrolled by medication;
11. Acute myocardial infarction based on clinical and/or electrocardiographic evidence;
12. Lung disease defined by a PaO2 ≤ 60mm Hg or an FiO2 ≥0.6;
13. Pregnancy as determined by βhCG results;
14. ≤2 weeks postpartum;
15. Eligible for an open ELAD clinical trial

Ages: 10 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult